CLINICAL TRIAL: NCT00605696
Title: Early Insulin Therapy and Development of Acute Respiratory Distress Syndrome
Brief Title: Early Insulin and Development of ARDS
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Albert Einstein College of Medicine (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Principal Investigator, Michelle Gong, Associate Professor, Albert Einstein College of Medicine
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 2009-462; R01HL086667 (NIH)
Record Dates: First submitted 2008-01-18; First posted 2008-01-31 (Estimated); Results first posted 2017-04-10 (Actual); Last update posted 2018-05-07 (Actual); Status verified 2018-04

CONDITIONS: Respiratory Distress Syndrome, Adult; Sepsis; Hyperglycemia
Keywords: Acute Respiratory Distress Syndrome; Acute Lung Injury
MeSH Terms: conditions — Respiratory Distress Syndrome; Sepsis; Hyperglycemia; Acute Lung Injury | interventions — Insulin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Experimental): Participants will receive insulin to target glucose 80-110 mg/dl within 6-12 hours after presenting to ED.
  Interventions: Drug: Insulin
- 2 (Active Comparator): Participants will receive insulin to target 150-180 mg/dl for 48 hours after ICU admission followed by usual clinical care.
  Interventions: Drug: Insulin

INTERVENTIONS:
Drug: Insulin — Participants will receive intravenous insulin to target tight glycemic control (80 to 110 mg/dL) for up to 48 hours after ICU admission.

SUMMARY:
Acute Lung Injury/Acute Respiratory Distress Syndrome (ALI/ARDS) is a severe lung condition that causes respiratory failure. Symptoms usually develop within 24 to 48 hours of an original injury or illness, and people with ALI/ARDS typically require care in the intensive care unit (ICU). Little is known about how to prevent the onset of ALI/ARDS. The purpose of this study is to examine if early infusions of insulin, known as intensive insulin therapy (IIT), can help prevent ALI/ARDS in hospitalized patients with high levels of blood sugars and severe infections.

DETAILED DESCRIPTION:
ALI/ARDS is a life-threatening condition that involves inflammation of the lungs and fluid accumulation in the air sacs, leading to low blood oxygen levels and respiratory failure. Common causes include pneumonia, lung trauma, and sepsis, a condition that can lead to widespread inflammation and blood clotting in response to an infection. Recent studies have shown that insulin, which is regularly used to control blood sugar levels, may prevent or lessen the risk of lung tissue inflammation and/or lung injury related to sepsis. Research has shown that critically ill ICU patients often benefit from receiving insulin to target 80-110 mg/dl , but it is not known if insulin to target these levels can prevent the onset of ALI/ARDS. Therapies to prevent ALI/ARDS should occur early, preferably even prior to ICU admission, because at least 38% of people with ALI/ARDS are diagnosed with the condition once they reach the ICU. The purpose of this study is to determine whether insulin to target 80-110 mg/dl administered to critically ill patients in the emergency department (ED) is more beneficial at preventing ALI/ARDS than insulin to target 150-180 mg/dl after ICU admission.

This study will enroll people who are hospitalized with high blood sugar levels and severe sepsis. Participants will be randomly assigned to receive IIT within 6-12 hours of ED presentation to target 80-110 mg/dl or target 150-180 mg/dl for 48 hours after admission to the ICU followed by usual care. Prior to ICU admission and 1, 3, and 7 days after ICU admission, blood will be collected and analyzed for markers of inflammation and lung injury. Blood samples will be stored for future research studies. While participants are in the hospital, their medical records will be reviewed to gather information on medical and family history, demographics, vital signs, laboratory test results, x-ray findings, and lung function. Study researchers will also monitor participants for the development of severe lung failure or other organ failures.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with severe sepsis, which is defined as sepsis AND one or more signs of organ dysfunction or hypotension
* Hyperglycemia (i.e., glucose level greater than 130 mg/dL on one or more tests)

Exclusion Criteria:

* Diabetic ketoacidosis
* Severe chronic liver disease with Child-Pugh score greater than 10 (Class C)
* Documented episodes of blood or plasma glucose less than 60 mg/dL within 24 hours of study entry
* Lack of any available IV access for insulin infusion
* Pregnant
* Known advanced directives against intubation or aggressive ICU care
* Inability to be enrolled into the study in the 12 hours following admission to the ED

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2008-04; Primary Completion 2011-12 (Actual); Study Completion 2013-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michelle Ng Gong, MD, MS, Principal Investigator — Montefiore Medical Center
Locations (1):
- Montefiore Medical Center, The Bronx, New York, United States

IPD SHARING:
Plan to Share IPD: Undecided

RESULTS

PARTICIPANT FLOW:
Groups:
- Early Insulin Group: Participants will receive insulin to target glucose of 80-110 mg/dl within 6-12 hours after presenting to ED for up to 48 hours after admission to the ICU.
- Control Group: Participants will receive insulin to target 150-180 mg/dl for 48 hours after ICU admission.
Period: Overall Study
Arm/Group | Early Insulin Group | Control Group
Started | 7 | 11
Completed | 7 | 11
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Early Insulin Group: Participants will receive IIT within 6-12 hours after presenting to ED.
  Insulin : Participants will receive intravenous insulin to target tight glycemic control (80 to 110 mg/dL) either in the ED or 48 hours after admission to the ICU.
- Control Group: Participants will receive insulin to target 150-180 mg/dl for 48 hours after ICU admission followed by usual clinical care.
  Insulin : Participants will receive intravenous insulin to target tight glycemic control (80 to 110 mg/dL) either in the ED or 48 hours after admission to the ICU.
- Total: Total of all reporting groups
Arm/Group | Early Insulin Group | Control Group | Total
Number analyzed (Participants) | 7 | 11 | 18
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 2 | 4 | 6
  >=65 years | 5 | 7 | 12
Age, Continuous [Mean (Standard Deviation); unit: years] | 74 (21) | 70 (18) | 72 (19)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7 | 5 | 12
  Male | 0 | 6 | 6
Region of Enrollment [Number; unit: participants]
  United States | 7 | 11 | 18

OUTCOME MEASURES:

1. Primary Outcome: Plasma Levels of Free Fatty Acids, Tumor Necrosis Factor-α, Interleukin-6, and Von Willebrand Factor Antigen
Time Frame: Measured at Day 1, 3 and 7
Population: Although blood samples were collected, there were no bioassays perfomed and therefore no data were collected from any study participants.
Groups:
- Early Insulin Group: Participants will receive intravenous insulin to target tight glycemic control (80 to 110 mg/dL) in the ED and after ICU admission for up to 48 hours.
- Control Group: Participants will receive insulin to target 150-180 mg/dl for 48 hours after ICU admission followed by usual clinical care.
Arm/Group | Early Insulin Group | Control Group
Number analyzed (Participants) | 0 | 0

2. Secondary Outcome: Murray Lung Injury Score
Description: Murray Lung Injury Score is a continuous score that quantifies the severity of lung injury and consist of components related to severity of hypoxia, pulmonary compliance, peep, and radiologic abnormalities. The scores range between 0 - 4. The higher the score, the greater the degree and severity of lung injury. The scale runs from 0-4, with 0 being the minimum and 4 the maximum score.
Time Frame: Measured at Day 3
Population: Change in Murray Lung Injury score from Day 3 to Day 0 (baseline)
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Early Insulin Group | Control Group
Number analyzed (Participants) | 7 | 11
units on a scale | 0.333 (0.81) | 0.323 (1.03)

ADVERSE EVENTS:
Arm/Group | Early Insulin Group | Control Group
All-Cause Mortality (participants affected / at risk) | 0/7 | 0/11
Serious Adverse Events (participants affected / at risk) | 0/7 | 0/11
Other Adverse Events (participants affected / at risk) | 2/7 | 0/11
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Early Insulin Group (N=7) | Control Group (N=11)
Hypoglycemia (Endocrine disorders) | 2 (2) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No